CLINICAL TRIAL: NCT02464111
Title: Short Term Response of Breast Milk Micronutrient Concentrations to a Lipid Based Nutrient Supplement in Guatemalan Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other); Blum Center for Developing Economies (Unknown); Fogarty International Center of the National Institute of Health (NIH); Center for the Studies of Sensory Impairment, Aging and Metabolism (CeSSIAM) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 723323-1; 5R25TW009343-03 (NIH)
Record Dates: First submitted 2015-04-22; First posted 2015-06-08 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Hypoxanthine Phosphoribosyltransferase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): Treatment 1: Control - no supplement given Treatment 2: Bolus - LNS supplement provided in one dose Treatment 3: Divided Dose - LNS supplement provided in 3 doses
  Interventions: Other: Treatment 1: Control; Dietary Supplement: Treatment 2: Bolus (LNS); Dietary Supplement: Treatment 3: Divided Dose (LNS)
- Group 2 (Experimental): Treatment 1: Control - no supplement given Treatment 3: Divided Dose - LNS supplement provided in 3 doses Treatment 2: Bolus - LNS supplement provided in one dose
  Interventions: Other: Treatment 1: Control; Dietary Supplement: Treatment 2: Bolus (LNS); Dietary Supplement: Treatment 3: Divided Dose (LNS)
- Group 3 (Experimental): Treatment 2: Bolus - LNS supplement provided in one dose Treatment 1: Control - no supplement given Treatment 3: Divided Dose - LNS supplement provided in 3 doses
  Interventions: Other: Treatment 1: Control; Dietary Supplement: Treatment 2: Bolus (LNS); Dietary Supplement: Treatment 3: Divided Dose (LNS)
- Group 4 (Experimental): Treatment 2: Bolus - LNS supplement provided in one dose Treatment 3: Divided Dose - LNS supplement provided in 3 doses Treatment 1: Control - no supplement given
  Interventions: Other: Treatment 1: Control; Dietary Supplement: Treatment 2: Bolus (LNS); Dietary Supplement: Treatment 3: Divided Dose (LNS)
- Group 5 (Experimental): Treatment 3: Divided Dose - LNS supplement provided in 3 doses Treatment 2: Bolus - LNS supplement provided in one dose Treatment 1: Control - no supplement given
  Interventions: Other: Treatment 1: Control; Dietary Supplement: Treatment 2: Bolus (LNS); Dietary Supplement: Treatment 3: Divided Dose (LNS)
- Group 6 (Experimental): Treatment 3: Divided Dose - LNS supplement provided in 3 doses Treatment 1: Control - no supplement given Treatment 2: Bolus - LNS supplement provided in one dose
  Interventions: Other: Treatment 1: Control; Dietary Supplement: Treatment 2: Bolus (LNS); Dietary Supplement: Treatment 3: Divided Dose (LNS)

INTERVENTIONS:
Other: Treatment 1: Control — No supplement provided.
Dietary Supplement: Treatment 2: Bolus (LNS) — One LNS supplement provided in a single bolus dose in the morning
Dietary Supplement: Treatment 3: Divided Dose (LNS) — One LNS supplement provided in 3 separate portions throughout the study visit

SUMMARY:
Research goals include evaluating the relative impact of maternal nutritional status versus recent dietary intake on breast milk micronutrient composition, and evaluating the impact of a maternal lipid based nutrient supplement (LNS) on breast milk micronutrient composition.

DETAILED DESCRIPTION:
The study includes a cross sectional and an interventional component. Maternal dietary intake and nutritional status will be compared to breast milk micronutrient composition in a cross sectional manner.

The short term effect of maternal dietary intake on breast milk micronutrient composition will be examined using an intervention with a controlled diet and LNS. Infants will be test-weighed during the LNS intervention in order to calculate the infant micronutrient intake from the control and LNS intervention days.

Mother-infant dyads will be recruited into the study and the order in which they will receive the 3 treatments will be randomized. All mothers will receive all treatments.

The mothers will be invited to the clinic on 4 separate occasions. During the first study visit, maternal blood will be collected, anthropometric indices will be assessed, and food frequency and demographic characteristic surveys will be administered. During the 2-4 visits, the LNS intervention will take place. Mothers will arrive at the clinic fasted, and a fasted milk collection will occur. Subsequently, mothers will be provided 3 meals based on local foods with low-nutrient density. Milk will be collected for 8 hours at each infant feed (ad libitum). A 24 hour dietary recall will be conducted. Mothers will receive 1) no LNS, 2) A single dose of LNS with breakfast, or 3) A single dose of LNS split into 3 parts with their meals throughout the day. Infants will be test weighed before and after each feed to calculate their nutrient intake from breast milk and the impact of the different supplementation schemes on their nutrient intake.

ELIGIBILITY:
Inclusion Criteria:

* Mother 18-40 years of age
* Apparently healthy, with no acute illness
* Willing to stay in clinic for breast milk sampling, and adhere to all study procedures
* 4-6 months of lactation and ≥ 8 breast feeding episodes per day (usual frequency is >20 times/day)
* Last birth was a singleton birth
* Only breastfeeding one child
* Child is 4-6 months of age

Exclusion Criteria:

* Current supplement use (iron + folic acid excepted)
* Self reported mastitis or other breast infections
* Reported problems with breastfeeding which might affect study procedures
* Last birth was premature (>4 weeks pre-term by maternal report)
* Measured body mass index (BMI) of less than 18.5 or a measured mid upper arm circumference (MUAC) of less than 12.5 cm
* Temporary- if the mother or her infant present with an acute illness, (for example flu or diarrhea,) they will be rescheduled to return on a later date when both are apparently healthy.
* Allergy to milk, milk products, or peanuts.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Cobalamin (vitamin B12) in Breast Milk | Breast milk cobalamin will be assessed in an 8-hour milk sample on each of three study visit days (Visits 2, 3, and 4.) Study visits/weeks 2, 3, & 4 will each be held approximately 1 week apart.
  We are observing the change in breast milk vitamin B12 over the course of 8 hours.
Change in Pyridoxal (vitamin B6) in Breast Milk | Breast milk pyridoxal will be assessed in an 8-hour milk sample on each of three study visit days (Visits 2, 3, and 4.) Study visits/weeks 2, 3, & 4 will each be held approximately 1 week apart.
  We are observing the change in breast milk vitamin B6 over the course of 8 hours.
Change in Riboflavin (vitamin B2) in Breast Milk | Breast milk riboflavin will be assessed in an 8-hour milk sample on each of three study visit days (Visits 2, 3, and 4.) Study visits 2, 3, & 4 will each be held approximately 1 week apart.
  We are observing the change in breast milk vitamin B2 over the course of 8 hours.
Change in Niacin (vitamin B3) in Breast Milk | Breast milk niacin will be assessed in an 8-hour milk sample on each of three study visit days (Visits 2, 3, and 4.) Study visits 2, 3, & 4 will each be held approximately 1 week apart.
  We are observing the change in breast milk vitamin B5 over the course of 8 hours.
Change in Thiamin (vitamin B1) in Breast Milk | Breast milk thiamin will be assessed in an 8-hour milk sample on each of three study visit days (Visits/weeks 2, 3, and 4.) Study visits 2, 3, & 4 will each be held approximately 1 week apart.
  We are observing the change in breast milk vitamin B1 over the course of 8 hours.

SECONDARY OUTCOMES:
Maternal cobalamin (vitamin B12) status | Measured once prior to first study visit (week 1)
  Maternal cobalamin (vitamin B12) status will be measured in blood.
Maternal pyridoxal (vitamin B6) status | Measured once prior to first study visit (week 1)
  Maternal pyridoxal (vitamin B6) will be measured in blood.
Maternal riboflavin (vitamin B2) status | Measured once prior to first study visit (week 1)
  Maternal riboflavin (vitamin B2) will be measured in blood.
Maternal niacin (vitamin B3) status | Measured once prior to first study visit (week 1)
  Maternal niacin (vitamin B5) will be measured in blood.
Maternal thiamin (vitamin B1) status | Measured once prior to first study visit (week 1)
  Maternal thiamin (vitamin B1) will be measured in blood.
Change in Infant Milk Consumption | Breast milk consumption for an 8-hour period will be assessed on each of three study visit days (Visits/weeks 2, 3, and 4). Study visits 2, 3, & 4 will each be held approximately 1 week apart.
  Infants will be test-weighed before and after each feed to calculate milk intake during the study visits. We are observing the change in breast milk intake over the course of 8 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana A Haber, B.S., Principal Investigator — USDA WHNRC, UC Davis
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Derived] Donohue JA, Solomons NW, Hampel D, Shahab-Ferdows S, Orozco MN, Allen LH. Micronutrient supplementation of lactating Guatemalan women acutely increases infants' intake of riboflavin, thiamin, pyridoxal, and cobalamin, but not niacin, in a randomized crossover trial. Am J Clin Nutr. 2020 Sep 1;112(3):669-682. doi: 10.1093/ajcn/nqaa147. PMID 32649760